CLINICAL TRIAL: NCT00094809
Title: Chemotherapy Administered Every 2 Weeks With or Without a Single Injection of Pegfilgrastim as First or Second-Line Treatment in Subjects With Locally Advanced or Metastatic Colon Cancer
Brief Title: Chemotherapy Administered Every 2 Weeks With or Without Pegfilgrastim in Subjects With Advanced or Metastatic Colon Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20020715; NCT00119327 (obsolete NCT alias)
Record Dates: First submitted 2004-10-26; First posted 2004-10-26 (Estimated); Results first posted 2011-01-06 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-09

CONDITIONS: Colon Cancer; Colorectal Cancer; Rectal Cancer
Keywords: Neulasta®; pegfilgrastim; Advanced; Chemotherapy
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms; Rectal Neoplasms | interventions — pegfilgrastim

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Pegfilgrastim (Active Comparator): 6 mg pegfilgrastim
  Interventions: Drug: Pegfilgrastim
- Placebo (Placebo Comparator): 6 mg placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Subjects randomized to placebo will receive a 6 mg subcutaneous injection once per cycle at least 24 hours after completion of 5-FU chemotherapy infusion. Subjects will continue to receive one injection per cycle until completion of 4 cycles, or until early termination from the study treatment period, whichever occurs first.
  Arms: Placebo
Drug: Pegfilgrastim — Subjects randomized to pegfilgrastim will receive a 6 mg subcutaneous injection once per cycle at least 24 hours after completion of 5-FU chemotherapy infusion. Subjects will continue to receive one injection per cycle until completion of 4 cycles, or until early termination from the study treatment period, whichever occurs first.
  Arms: Pegfilgrastim

SUMMARY:
The purpose of this research study is to evaluate the safety and effectiveness of pegfilgrastim in reducing grade 3/4 neutropenia when given after one of three chemotherapy regimens (FOIL, FOLFOX or FOLFIRI) in patients with locally advanced or metastatic colorectal cancer. This study is considered to be "investigational" because the time between receiving pegfilgrastim and the next cycle of chemotherapy is only 11 days.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic colorectal adenocarcinoma not curable by surgery or amenable to radiation therapy with curative intent.
* Histologically or cytologically documented locally advanced or metastatic colorectal cancer. The site of the primary lesion must be or has been confirmed endoscopically, radiologically, or surgically to be or has been in the large bowel.
* Measurable or evaluable disease.
* ECOG performance status 0, 1 or 2
* Life expectancy ≥ 12 weeks
* All of the following: (1) ≥ 4 weeks must have elapsed from the time of major surgery and subjects must have recovered from the effects (e.g., laparotomy); (2) ≥ 2 weeks must have elapsed from the time of minor surgery and subjects must have recovered from the operation (insertion of a vascular access device is not considered major or minor surgery); (3) ≥ 4 weeks must have elapsed from the time of major radiotherapy (e.g., chest or bone palliative radiation therapy).
* Subjects may have received prior adjuvant therapy and one prior chemotherapy regimen for metastatic disease providing 30 days has elapsed from last chemotherapy dose.
* Subject must have recovered from prior chemotherapy complications and in the opinion of the investigator, the subjects current status does not place the subject at risk for entry into the trial.
* Subjects with prior exposure to both oxaliplatin and irinotecan will not be eligible to participate in this study. However, if subject received prior therapy with oxaliplatin, they will be eligible to receive the FOLFIRI regimen. If subject received prior therapy with irinotecan, they will be eligible to receive the FOLFOX regimen.
* Age ≥ 18 years
* Absolute neutrophil count ≥ 1.5 x 109/L
* Platelet count ≥100 x 109/L
* Hemoglobin ≥ 9.0 g/dL (subjects may be receive a red blood cell transfusion to achieve this requirement)
* Creatinine ≤ 1.5 x UNL
* Total bilirubin ≤ 1.5 mg/dL (≤ 25.65 μmol/L), regardless of whether subjects have liver involvement secondary to tumor
* Aspartate aminotransferase ≤ 5 x UNL
* Alkaline phosphatase ≤ 5 x UNL
* Informed consent to participate on the study.

Exclusion Criteria:

* Standard chemoradiation as adjuvant treatment for colorectal cancer will be allowed, but prior radiotherapy to >15% of bone marrow or outside of standard adjuvant colorectal cancer chemoradiation is not allowed.
* Known central nervous system metastases or carcinomatous meningitis.
* Predisposing colonic or small bowel disorders in which the symptoms are uncontrolled as indicated by baseline pattern of >3 loose stools daily in subjects without a colostomy or ileostomy. Subjects with a colostomy or ileostomy may be entered at the Investigator's discretion.
* Pleural effusion or ascites, which cause respiratory compromise (≥Grade 2 dyspnea).
* Concurrent use of other investigational agents.
* No active infection requiring the start of systemic (intravenous or oral) anti-infective (antibiotic, antifungal, antiviral) within 72 hours of the administration of the first cycle of study chemotherapy.
* Symptomatic sensory peripheral neuropathy.
* The following conditions: Uncontrolled high blood pressure; unstable angina; symptomatic congestive heart failure; myocardial infarction ≤ 6 months prior to randomization; serious uncontrolled cardiac arrhythmia; New York Heart Association classification III or IV.
* Prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, adequately treated noninvasive carcinomas, or other cancer from which the patient has been disease-free for at least five years.
* Interstitial pneumonia or extensive and symptomatic interstitial fibrosis of the lung.
* Medical or psychiatric conditions which, in the opinion of the Investigator, make participation in an investigational trial of this nature a poor risk.
* Known sensitivity to E. coli derived products (e.g., Filgrastim, HUMULIN® insulin, L-asparaginase, HUMATROPE® Growth Hormone, INTRON® A) or known sensitivity to any of the products to be administered during dosing.
* Subject is currently enrolled or has not yet completed at least 30 days since ending other investigational device or drug trial(s) or is receiving other investigational agent(s).
* Subject of child-bearing potential is evidently pregnant (e.g., positive HCG test) or is breast feeding.
* Subject is not using adequate contraceptive precautions.
* Subject will not be available for follow-up assessment.
* Concerns for subject's compliance with the protocol procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2003-02-01 (Actual); Primary Completion 2006-05-19 (Actual); Study Completion 2008-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Hecht JR, Pillai M, Gollard R, Heim W, Swan F, Patel R, Dreiling L, Mo M, Malik I. A randomized, placebo-controlled phase ii study evaluating the reduction of neutropenia and febrile neutropenia in patients with colorectal cancer receiving pegfilgrastim with every-2-week chemotherapy. Clin Colorectal Cancer. 2010 Apr;9(2):95-101. doi: 10.3816/CCC.2010.n.013. PMID 20378503
- [Derived] Lyman GH, Reiner M, Morrow PK, Crawford J. The effect of filgrastim or pegfilgrastim on survival outcomes of patients with cancer receiving myelosuppressive chemotherapy. Ann Oncol. 2015 Jul;26(7):1452-8. doi: 10.1093/annonc/mdv174. Epub 2015 Apr 7. PMID 25851633
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: FDA-approved Drug Labeling — http://www.neulasta.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 12 February 2003 through 13 January 2006
Groups:
- Pegfilgrastim (Neulasta): Pegfilgrastim 6 mg by subcutaneous injection once every 2 weeks at least 24 hours after 5-fluorouracil infusion
- Placebo: Placebo administered by subcutaneous injection once every 2 weeks at least 24 hours after 5-fluorouracil infusion
Period: Overall Study
Arm/Group | Pegfilgrastim (Neulasta) | Placebo
Started | 126 | 126
Received Study Drug | 124 | 118
Properly Consented; Received Study Drug | 123 | 118
Completed All 4 Cycles of Treatment | 98 | 90
Completed | 74 (Subjects who completed treatment and Long term follow up (LTFU)) | 61 (Subjects who completed treatment and LTFU)
Not Completed | 52 | 65
Not completed — Protocol deviation | 2 | 2
Not completed — Noncompliance | 1 | 0
Not completed — Adverse Event | 3 | 1
Not completed — Withdrawal by Subject | 8 | 9
Not completed — Disease progression | 3 | 3
Not completed — Physician Decision | 3 | 5
Not completed — Lost to Follow-up | 6 | 6
Not completed — Death | 19 | 25
Not completed — Protocol-specified criteria | 1 | 1
Not completed — Other | 2 | 4
Not completed — Informed consent signed after treatment | 1 | 0
Not completed — Study drug not received | 2 | 8
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pegfilgrastim (Neulasta) | Placebo | Total
Number analyzed (Participants) | 123 | 118 | 241
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.4 (12.26) | 62.9 (13.21) | 62.7 (12.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 34 | 79
  Male | 78 | 84 | 162
Race/Ethnicity, Customized [Number; unit: Participants]
  White or Caucasian | 103 | 84 | 187
  Black or African American | 12 | 12 | 24
  Hispanic or Latino | 3 | 16 | 19
  Asian | 3 | 3 | 6
  Japanese | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 3 | 3
  Other | 1 | 0 | 1
Chemotherapy Regimen [Number; unit: Participants] — FOIL = 5-fluorouracil, oxaliplatin, irinotecan, and leucovorin; FOLFOX = 5-fluorouracil, oxaliplatin, and leucovorin; FOLFIRI = 5-fluorouracil, irinotecan, and leucovorin
  Participants
    FOIL | 30 | 30 | 60
    FOLFOX | 61 | 58 | 119
    FOLFIRI | 32 | 30 | 62

OUTCOME MEASURES:

1. Primary Outcome: Grade 3 or 4 Neutropenia
Description: Grade 3 or 4 neutropenia, defined as an absolute neutrophil count (ANC) < 1 x 10^9/L, in any of the first four cycles of treatment
Time Frame: First 4 cycles of treatment (8 weeks)
Population: Primary Analysis Set, composed of all participants who received study drug and who signed an informed consent before any invasive procedures
Measure: Number; unit: Participants
Arm/Group | Pegfilgrastim (Neulasta) | Placebo
Number analyzed (Participants) | 123 | 118
Participants | 16 | 51
Statistical Analysis 1: Comparison: Pegfilgrastim (Neulasta) vs Placebo; Test type: Superiority or Other; p < 0.0001, Mantel Haenszel; Adjusted for chemotherapy regimen; Odds Ratio (OR) = 0.19, 95% CI [0.10 to 0.37] — Common odds ratio of the pegfilgrastim group compared to the placebo group

2. Secondary Outcome: Dose Delay or Reduction Due to Neutropenia
Description: Dose delay or reduction in chemotherapy doses due to neutropenia
Time Frame: First 4 cycles of treatment (8 weeks)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Pegfilgrastim (Neulasta) | Placebo
Number analyzed (Participants) | 123 | 118
Participants | 5 | 26
Statistical Analysis 1: Comparison: Pegfilgrastim (Neulasta) vs Placebo; Test type: Superiority or Other; p < 0.0001, Mantel Haenszel; Adjusted for chemotherapy regimen; Treatment difference = -18, 95% CI [-26.2 to -9.8] — Treatment difference in percentage of participants (pegfilgrastim group - placebo group)

3. Secondary Outcome: Dose Delay or Reduction for Any Reason
Description: Dose delay or reduction in chemotherapy dose during the first 4 cycles for any reason
Time Frame: First 4 cycles of treatment (8 weeks)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Pegfilgrastim (Neulasta) | Placebo
Number analyzed (Participants) | 123 | 118
Participants | 41 | 53
Statistical Analysis 1: Comparison: Pegfilgrastim (Neulasta) vs Placebo; Test type: Superiority or Other; p = 0.0646, Mantel Haenszel; Adjusted for chemotherapy regimen; Treatment difference = -12, 95% CI [-23.7 to 0.5] — Treatment difference in percentage of participants (pegfilgrastim group - placebo group)

4. Secondary Outcome: Febrile Neutropenia
Description: Febrile neutropenia, Defined as a temperature ≥ 38.2 °C on a given day, with an ANC < 1.0 x 10^9/L recorded on the same day or the next day, during any of the first 4 cycles of treatment.
Time Frame: First 4 cycles of treatment (8 weeks)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Pegfilgrastim (Neulasta) | Placebo
Number analyzed (Participants) | 123 | 118
Participants | 3 | 10
Statistical Analysis 1: Comparison: Pegfilgrastim (Neulasta) vs Placebo; Test type: Superiority or Other; p = 0.0384, Mantel Haenszel; Adjusted for chemotherapy regimen; Odds Ratio (OR) = 0.27, 95% CI [0.07 to 1.00] — Common odds ratio of pegfilgrastim group compared to placebo group

5. Secondary Outcome: Hospitalization Due to a Neutropenia-Related Event
Description: Hospitalization because of a neutropenia-related event during the first 4 cycles of treatment
Time Frame: First 4 cycles of neutropenia (8 weeks)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Pegfilgrastim (Neulasta) | Placebo
Number analyzed (Participants) | 123 | 118
Participants | 7 | 9
Statistical Analysis 1: Comparison: Pegfilgrastim (Neulasta) vs Placebo; Test type: Superiority or Other; p = 0.5514, Mantel Haenszel; Adjusted for chemotherapy regimen; Odds Ratio (OR) = 0.73, 95% CI [0.26 to 2.04] — Common odds ratio for pegfilgrastim group compared to placebo group

6. Secondary Outcome: Progression-Free Survival
Description: Kaplan-Meier estimate of the median time to disease progression or death
Time Frame: Up to 24 months after first four cycles of treatment
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Pegfilgrastim (Neulasta) | Placebo
Number analyzed (Participants) | 123 | 118
Days | 318 [258 to 387] | 322 [268 to 387]

7. Secondary Outcome: Objective Tumor Response
Description: Objective tumor response (complete or partial) at the end of treatment, defined as a reduction of at least 50% in the area of all measurable lesions (partial response) or disappearance of all measurable or evaluable disease without the development of new lesions (complete response) on computed tomographic (CT) or other scanning.
Time Frame: First 4 cycles of treatment (8 weeks)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Pegfilgrastim (Neulasta) | Placebo
Number analyzed (Participants) | 123 | 118
Participants | 34 | 37
Statistical Analysis 1: Comparison: Pegfilgrastim (Neulasta) vs Placebo; Test type: Superiority or Other; p = 0.5434, Mantel Haenszel; Adjusted for chemotherapy regimen; Treatment difference = -3.5, 95% CI [-14.8 to 7.8] — Treatment difference (pegfilgrastim group - placebo group) in the percentage of participants with a complete or partial response

8. Secondary Outcome: Survival
Description: Death from any cause through the end of the follow-up period
Time Frame: Up to 24 months after first four cycles of treatment
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Pegfilgrastim (Neulasta) | Placebo
Number analyzed (Participants) | 123 | 118
Participants | 47 | 49
Statistical Analysis 1: Comparison: Pegfilgrastim (Neulasta) vs Placebo; Test type: Superiority or Other; Treatment difference = -12.1, 95% CI [-28.1 to 4.0] — Kaplan-Meier estimates of the difference in percent mortality for the pegfilgrastim group - placebo group. Median survival time was not reached for the pegfilgrastim group

9. Secondary Outcome: Antibiotic Use Due to Febrile Neutropenia
Description: Antibiotic use during any of the first 4 cycles of treatment due to febrile neutropenia.
Time Frame: First 4 cycles of treatment (8 weeks)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Pegfilgrastim (Neulasta) | Placebo
Number analyzed (Participants) | 123 | 118
Participants | 2 | 8
Statistical Analysis 1: Comparison: Pegfilgrastim (Neulasta) vs Placebo; Test type: Superiority or Other; p = 0.0457, Mantel Haenszel; Adjusted for chemotherapy regimen; Odds Ratio (OR) = 0.23, 95% CI [0.05 to 1.09] — Common odds ratio for pegfilgrastim group compared to placebo group

10. Primary Outcome: Grade 4 Neutropenia
Description: Grade 4 neutropenia, defined as an absolute neutrophil count (ANC) <0.5 x 10^9/L, in any of the first four cycles of treatment
Time Frame: First 4 cycles of treatment (8 weeks)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Pegfilgrastim (Neulasta) | Placebo
Number analyzed (Participants) | 123 | 118
Participants | 13 | 17
Statistical Analysis 1: Comparison: Pegfilgrastim (Neulasta) vs Placebo; Test type: Superiority or Other; p = 0.3792, Mantel Haenszel; Adjusted for chemotherapy regimen; Odds Ratio (OR) = 0.71, 95% CI [0.32 to 1.53] — Common odds ratio of the pegfilgrastim group compared to the placebo group

ADVERSE EVENTS:
Time Frame: During treatment period and including 30 days after last dose of IP
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
  One subject randomized to pegfilgrastim arm was not summarized in the safety analysis set due to improper informed consent.
  Another subject who was randomized to placebo arm but received pegfilgrastim and was summarized in pegfilgrastim arm.
Arm/Group | Placebo | Pegfilgrastim
Serious Adverse Events (participants affected / at risk) | 36/117 | 44/124
Other Adverse Events (participants affected / at risk) | 108/117 | 112/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=117) | Pegfilgrastim (N=124)
Agranulocytosis (Blood and lymphatic system disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 6 | 3
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 7
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1
Colon gangrene (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 7
Faecal incontinence (Gastrointestinal disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 7 | 2
Proctalgia (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 6 | 2
Asthenia (General disorders) | 0 | 1
Chest pain (General disorders) | 2 | 0
Disease progression (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 3
Abdominal abscess (Infections and infestations) | 0 | 1
Catheter sepsis (Infections and infestations) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 2
Gastrointestinal infection (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 1
Peritonitis bacterial (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 5
Sepsis (Infections and infestations) | 1 | 2
Septic shock (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 1
Wound infection staphylococcal (Infections and infestations) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Intestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 1
Post procedural diarrhoea (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Antimicrobial susceptibility test resistant (Investigations) | 0 | 1
Blood culture positive (Investigations) | 0 | 1
Prothrombin level increased (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 6 | 14
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Dysarthria (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 2 | 0
Renal failure (Renal and urinary disorders) | 1 | 1
Ureteric obstruction (Renal and urinary disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive airways disease exacerbated (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Deep vein thrombosis (Vascular disorders) | 3 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=117) | Pegfilgrastim (N=124)
Anaemia (Blood and lymphatic system disorders) | 32 | 36
Leukocytosis (Blood and lymphatic system disorders) | 3 | 7
Neutropenia (Blood and lymphatic system disorders) | 55 | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 9 | 9
Abdominal distension (Gastrointestinal disorders) | 0 | 7
Abdominal pain (Gastrointestinal disorders) | 16 | 22
Abdominal pain upper (Gastrointestinal disorders) | 2 | 8
Constipation (Gastrointestinal disorders) | 13 | 14
Diarrhoea (Gastrointestinal disorders) | 53 | 62
Dyspepsia (Gastrointestinal disorders) | 3 | 7
Mouth ulceration (Gastrointestinal disorders) | 4 | 7
Nausea (Gastrointestinal disorders) | 53 | 69
Stomatitis (Gastrointestinal disorders) | 8 | 8
Vomiting (Gastrointestinal disorders) | 22 | 35
Asthenia (General disorders) | 6 | 22
Chest pain (General disorders) | 2 | 8
Fatigue (General disorders) | 44 | 49
Mucosal inflammation (General disorders) | 6 | 8
Oedema peripheral (General disorders) | 6 | 8
Pain (General disorders) | 14 | 8
Pyrexia (General disorders) | 9 | 18
Weight decreased (Investigations) | 8 | 19
Anorexia (Metabolism and nutrition disorders) | 14 | 29
Decreased appetite (Metabolism and nutrition disorders) | 4 | 10
Dehydration (Metabolism and nutrition disorders) | 10 | 14
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 18
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 10
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 13
Dizziness (Nervous system disorders) | 5 | 8
Headache (Nervous system disorders) | 7 | 9
Hypoaesthesia (Nervous system disorders) | 7 | 8
Neuropathy (Nervous system disorders) | 5 | 8
Neuropathy peripheral (Nervous system disorders) | 3 | 7
Paraesthesia (Nervous system disorders) | 5 | 10
Anxiety (Psychiatric disorders) | 6 | 4
Depression (Psychiatric disorders) | 4 | 9
Insomnia (Psychiatric disorders) | 9 | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 12
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 | 6
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 8
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 15
Rash (Skin and subcutaneous tissue disorders) | 6 | 5
Hypotension (Vascular disorders) | 2 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multi-center studies, the investigator agrees not to publish any results before the first multi-center publication.